CLINICAL TRIAL: NCT01501786
Title: The Effect of Small-dose Ketamine on Depression of Respiratory and Cardiac Functions Caused by Propofol in Pediatric Cardiac Catheterization
Brief Title: Does Ketamine Attenuate Depression of Respiratory and Cardiac Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibaraki Children's Hospital (Other)
Responsible Party: Principal Investigator, Kazuhiko Okuyama, MD, Head of Anesthesiology department, Ibaraki Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: ketamine in sedation
Record Dates: First submitted 2011-12-10; First posted 2011-12-29 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Congenital Heart Disease; Sedated for Cardiac Catheterization
Keywords: children; sedation; propofol; ketamine
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Sodium Chloride; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- control (Sham Comparator): propofol and saline are administered
  Interventions: Drug: control
- Ket10 (Experimental): ketamine is co-administered with propofol
  Interventions: Drug: Ket10
- Ket20 (Experimental): ketamine is co-administered with porpofol
  Interventions: Drug: Ket20

INTERVENTIONS:
Drug: control — propofol 8mg/kg/h saline 0.24 ml/kg/h
  Other Names: saline with propofol
  Arms: control
Drug: Ket10 — propofol 6.4 mg/kg/h ketamine 10 microg/kg/min
  Other Names: ketamine 10 γ
  Arms: Ket10
Drug: Ket20 — propofol 4.8 mg/kg/h ketamine 20 microg/kg/min
  Other Names: ketamine 20 γ
  Arms: Ket20

SUMMARY:
Normal cardiac and respiratory functions should be maintained during pediatric cardiac catheterization. Propofol has become a popular choice for sedation in children, however, it depresses cardiac and respiratory functions. Some investigators reported that ketamine attenuates its depressant effect, but it remains unclear whether ketamine reduces cardiac and respiratory depression caused by propofol in pediatric cardiac catheterization.

ELIGIBILITY:
Inclusion Criteria:

* 7kg-25kg (6mo-10yrs) children who undergo cardiac catheterization

Exclusion Criteria:

* patients who have neurological disease,
* endocrinological disease,
* airway anomaly, who require positive pressure ventilation

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
difference of end tidal partial pressure of carbon dioxide between the groups | 30 and 60 min after anesthetic induction
difference of partial pressure of arterial carbon dioxide between the groups | 60 min after anesthetic induction on average
heart rate change from baseline value | 30 and 60 min after anesthetic induction
non-invasive blood pressure change from baseline value | 30 and 60 min after anesthetic induction

SECONDARY OUTCOMES:
movement at topical anesthetic injection | 20 min after anesthetic induction on average
  1. none (no movement or slight movement unnecessary to restrain)
  2. mild (movement necessary to restrain, limited to lower extremities)
  3. moderate (strong movement of lower extremities and movement of upper extremities unvecessary to restrain)
  4. severe (movement necessary to restrain upper extremities and body trunk in addition to lower extremities, or some vacalization)
the number of times that secreted saliva is aspirated by an attending anesthesiologist | From anesthetic induction to termination of anethetics administration, which is not over 2 hours from anesthetic induction

CONTACTS AND LOCATIONS:
Overall Officials: Kazuhiko Okuyama, MD, Study Chair — Ibaraki Children's Hospital; Yuki Takeda, MD, Principal Investigator — Ibaraki Children's Hospital
Locations (1):
- Ibaraki Children's Hospital, Mito, Ibaraki, Japan